CLINICAL TRIAL: NCT02815670
Title: Single Dose, Open Label, Uncontrolled, Safety Trial of Intravenous Administration of Idarucizumab to Paediatric Patients Enrolled From Ongoing Phase IIb/III Clinical Trials With Dabigatran Etexilate for the Treatment and Secondary Prevention of Venous Thromboembolism.
Brief Title: Reversal Dabigatran Anticoagulant Effect With Idarucizumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1321.7; 2015-002177-37 (EudraCT Number)
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-03

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — idarucizumab

ARMS (1):
- Idarucizumab (Experimental)
  Interventions: Drug: Idarucizumab

INTERVENTIONS:
Drug: Idarucizumab

SUMMARY:
The trial objective is to demonstrate the safety of idarucizumab, as assessed by the occurence of patients with drug related adverse events (including immune reactions) and all-cause mortality in paediatric venous thromboembolism patients treated with dabigatran in ongoing clinical trials who require emergency surgery/urgent procedures or patients who have life-threatening or uncontrolled bleeding which requires urgent intervention, when rapid reversal of the anticoagulant effect of dabigatran is needed.

ELIGIBILITY:
Inclusion criteria:

Patients taking dabigatran etexilate in the paediatric trials 1160.106 or 1160.108 are eligible for this trial if they meet the following criteria:

Group A:

* Overt bleeding judged by the treating physician to require a reversal agent.
* Currently taking dabigatran etexilate in the context of a clinical trial with dabigatran etexilate (1160.106 or 1160.108).
* Male or female patients from 0 to less than 18 years of age at the time of informed consent/assent for participation in trial 1160.106 or in trial 1160.108.
* Female patients of childbearing potential (defined as having experienced menarche) must have followed the contraception requirements according to the dabigatran trial 1160.106 or trial 1160.108 in which they are enrolled.
* Written informed consent provided by the patient (and/or the patient's legally accepted representative) and assent provided by the patient (if applicable) at the time of informed consent signature in accordance with Good Clinical Practice (GCP) and local legislation prior to admission to the trial. If the child is unable to give assent at the time of the emergency, the assent, when applicable will be obtained as soon as feasible.

Group B:

* A condition requiring an emergency surgery or invasive procedure where adequate haemostasis is required. Emergency is defined as need for surgery or intervention within the following 8 hours.
* Currently taking dabigatran etexilate in the context of a clinical trial with dabigatran etexilate (1160.106 or 1160.108).
* Male or female patients from 0 to less than 18 years of age at the time of informed consent/assent for participation in trial 1160.106 or in trial 1160.108.
* Female patients of childbearing potential (defined as having experienced menarche) must have followed the contraception requirements according to the dabigatran trial 1160.106 or trial 1160.108 in which they are enrolled.
* Written informed consent provided by the patient (and/or the patient's legally accepted representative) and assent provided by the patient (if applicable) at the time of informed consent signature in accordance with GCP and local legislation prior to admission to the trial. If the child is unable to give assent at the time of the emergency, the assent, when applicable will be obtained as soon as feasible.

Exclusion criteria:

Group A:

* Patients with minor bleeding (e.g. epistaxis, haematuria) who can be managed with standard supportive care.
* Patients with no clinical signs of bleeding.
* Patients with body weight < 2.5 kg
* Contraindications to trial medication including known hypersensitivity to the drug or its excipients; i.e. patients with hereditary fructose intolerance who may react to sorbitol.
* Female patients who are pregnant, nursing, or who plan to become pregnant while in the trial.

Group B:

* A surgery or procedure which is elective or where the risk of uncontrolled or unmanageable bleeding is low.
* Patients with body weight < 2.5 kg
* Contraindications to trial medication including known hypersensitivity to the drug or its excipients; i.e. patients with hereditary fructose intolerance who may react to sorbitol.
* Female patients who are pregnant, nursing, or who plan to become pregnant while in the trial.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2019-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Russia (2):
  - Children Rep.Clin.Hosp of MoH,Cardio Vas.surgery Dept, Kazan, Kazan'
  - Regional Clin.Hosp.1,Congen.heart defects&child.Cardiol.dept, Tyumen

REFERENCES:
- [Derived] Albisetti M, Schlosser A, Brueckmann M, Gropper S, Glund S, Tartakovsky I, Brandao LR, Reilly PA. Rationale and design of a phase III safety trial of idarucizumab in children receiving dabigatran etexilate for venous thromboembolism. Res Pract Thromb Haemost. 2017 Nov 17;2(1):69-76. doi: 10.1002/rth2.12053. eCollection 2018 Jan. PMID 30046708
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, uncontrolled case series trial, with a single treatment arm of idarucizumab in patients with venous thromboembolism treated with dabigatran etexilate in ongoing Boehringer Ingelheim pediatric clinical trials (1160.106 and 1160.108). Treatment period was around 1 day followed by 29 days of safety follow-up period.
Pre-assignment Details: All subjects were screened for eligibility to participants in the trial. Subjects attended specialist sites which would then ensure that they met all strictly implemented inclusion/exclusion criteria. Subjects were not to be assigned to treatment groups if any one of the specific entry criteria were violated.
Groups:
- Idarucizumab: 2.5 gram (g) per 50 milliliter (mL) vial of Idarucizuma was administrated via intravenous injection (vial 1) with (in order of preference): a 5 minutes (min) infusion with an infusion pump, a 10 to 15 min drip, or intravenous push with a syringe followed by another injection (vial 2) of same dosage of Idarucizumab for participants who were treated with dabigatran and had uncontrolled or life threatening bleeding that required urgent medical or surgical intervention or who required emergency surgery/urgent procedures where adequate haemostasis was required (total dosage: up to 5g based on the weight of participant). Two equal injection parts were administered no more than 15 min apart. The time between start of injection of the first vial and end of the second vial was 22 min followed by 24 hours post-dose observation period.
Period: Overall Study
Arm/Group | Idarucizumab
Started | 1
Completed | 0
Not Completed | 1
Not completed — Prematurely discontinued of the trial | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): including all patients who received any dose of idarucizumab. The TS was used to assess safety, clinical endpoints, demographics and baseline characteristics, concomitant diagnosis/therapy and medical history, and antidrug antibodies (ADA).
Arm/Group | Idarucizumab
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | NA (NA) — Information were collected but not reported for protection of pediatric participant.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Information were collected but not reported for protection of pediatric participant.
  Male | NA — Information were collected but not reported for protection of pediatric participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants] | NA — Race and ethnicity were collected but not reported for protection of pediatric participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-related Adverse Events (AEs)
Description: Number of participants with drug-related adverse events (AEs) including immune reactions and all cause mortality during the trial.
Time Frame: From vial 1 of Idarucizumab until prematurely discontinued of the trial, up to 25 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Idarucizumab
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Percent Change of Coagulation Time for Diluted Thrombin Time (dTT) and Ecarin Clotting Time (ECT) at 30 Minutes Post-dose Compared With Pre-dose
Description: Percent change of coagulation time for diluted thrombin time (dTT) and ecarin clotting time (ECT) at 30 minutes (min) post-dose compared with pre-dose. Central blood sampling for dTT, ECT were to occur immediately prior to administration of each vial of Idarucizumab and post-dose at 30min, 4h, 12h and 24h.
Time Frame: At immediately prior to administration of vial 1 of Idarucizumab and 30 minutes (min) post vial 2 administration.
Population: Pharmacodynamic (PD) set (PDS): comprising all patients in the TS who provided at least 1 evaluable pre-dose and at least 1 post-dose observation for PD endpoints or biomarker measures. The PDS was used for the PD endpoint analyses. Note that for different PD endpoints or biomarkers, the number of evaluable patients could differ between endpoints.
Measure: Number; unit: Percentage of time in seconds
Arm/Group | Idarucizumab
Number analyzed (Participants) | 1
Percentage of time in seconds
  Diluted thrombin time (dTT) | -46.3
  Ecarin clotting time (ECT) | -67.8

3. Secondary Outcome: Time to Achieve Reversal of the Dabigatran Effect (Based on the Coagulation Time for dTT and ECT)
Description: Idarucizumab administration resulted in normalisation of dTT and ECT. Time to achieve reversal of anticoagulant effect of dabigatran based on the coagulation time for dTT and ECT, at any time point from the end of the second injection (vial 2) up to 24 hours (h). Reversal of the dabigatran effect at time t was defined as the 100 percent (%) *(pre-dose coagulation time - post-dose coagulation time at time t)/(pre-dose coagulation test - upper limit of normal).
  Values equal to or higher than 100% were interpreted as reversal. Central blood sampling for dTT, ECT were to occur immediately prior to administration of each vial of Idarucizumab and post-dose at 30min, 4h, 12h and 24h.
Time Frame: From end of vial 2 of Idarucizumab up to 24h.
Population: as for outcome 2
Measure: Number; unit: Minutes
Arm/Group | Idarucizumab
Number analyzed (Participants) | 1
Minutes | 30

4. Secondary Outcome: Duration of Reversal of the Dabigatran Effect Sustained up to 24 Hours Post-dose (Based on the Coagulation Time for dTT and ECT)
Description: Duration of reversal, defined as the time period a patient remained completely reversed based on dTT and ECT, up to 24 hours post-dose or restarting the treatment of anticoagulation. Central blood sampling for dTT, ECT were to occur immediately prior to administration of each vial of idarucizumab and post-dose at 30min, 4h, 12h and 24h.
Time Frame: From end of vial 2 of Idarucizumab up to 24h.
Population: as for outcome 2
Measure: Number; unit: Hours
Arm/Group | Idarucizumab
Number analyzed (Participants) | 1
Hours | 23.5

5. Secondary Outcome: Number of Participants With Cessation of Bleeding
Time Frame: From vial 1 of Idarucizumab through vial 2 of Idarucizumab, up to 24h 30min.
Population: Treated set (TS): including all patients who received any dose of Idarucizumab. The TS was used to assess safety, clinical endpoints, demographics and baseline characteristics, concomitant diagnosis/therapy and medical history, as well as ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Idarucizumab
Number analyzed (Participants) | 1
Participants | 1

6. Secondary Outcome: Number of Participants Per Bleeding Status During the Trial
Description: Numbers of participants whose bleeding had stopped, reduced, unchanged, worsened or not applicable during the trial were characterized.
Time Frame: From vial 1 of Idarucizumab until prematurely discontinued of the trial, up to 25 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Idarucizumab
Number analyzed (Participants) | 1
Participants
  Stopped | 1
  Reduced | 0
  Unchanged | 0
  Worsened | 0
  Not applicable | 0

7. Secondary Outcome: Number of Participants With Clinical Conditions Contributing to Bleeding During the Trial
Description: Number of participants with clinical conditions (trauma, surgery and use of antiplatelet) contributing to bleeding during the trial were characterized.
Time Frame: From vial 1 of Idarucizumab until prematurely discontinued of the trial, up to 25 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Idarucizumab
Number analyzed (Participants) | 1
Participants
  Trauma | 1
  Surgery | 0
  Use of antiplatelet | 0

8. Secondary Outcome: Number of Participants Developing Treatment-emergent Antidrug Antibodies (ADA) With Cross Reactivity to Idarucizumab
Time Frame: At day 25 post vial 2 of Idarucizumab administration, up to 1 day
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Idarucizumab
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: From vial 1 of Idarucizumab until prematurely discontinued of the trial, up to 25 days
Description: Treated set (TS): including all patients who received any dose of Idarucizumab. The TS was used to assess safety, clinical endpoints, demographics and baseline characteristics, concomitant diagnosis/therapy and medical history, and antidrug antibodies (ADA).
Arm/Group | Idarucizumab
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idarucizumab (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
The patient completed the treatment period, but the end-of-trial visit was by mistake scheduled 5 days earlier. Thus, the patient was formally considered as having prematurely discontinued the trial although all planned visits were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT02815670/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/70/NCT02815670/SAP_001.pdf